CLINICAL TRIAL: NCT05961462
Title: Effects of Exercise Training on Patients With Long COVID-19, a Single-center, Randomized, Controlled Study
Brief Title: Effects of Exercise Training on Patients With Long COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Huan Ma, Deputy Director of Cardiology, Director of the Department of Cardiac Rehabilitation, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2023-053-02
Record Dates: First submitted 2023-07-24; First posted 2023-07-27 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Long COVID-19
Keywords: Long COVID-19; Exercise training; Cardiopulmonary fitness; Symptom improvement
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training group (Active Comparator): Exercise training containing 12 sessions of a structured aerobic exercise training program over 4 weeks (3 times per week).
  Interventions: Behavioral: Exercise training
- Attention control (No Intervention): Conventional care.

INTERVENTIONS:
Behavioral: Exercise training — Patients randomized to the exercise group will be offered aerobic exercise plan containing 12 sessions over 4 weeks (3 times per week).
  Arms: Exercise training group

SUMMARY:
Effects of Exercise training on Patients With Long COVID-19, is a single-center, randomized, controlled trial designed to evaluate the effects of 4- week aerobic exercise administered to patients with long COVID-19 symptoms. The main outcome is cardiopulmonary fitness and long COVID-19 symptom improvement. Quality of life, depression, anxiety, insomnia status and perceived stress will also be assessed before and after the exercise program.

DETAILED DESCRIPTION:
Long COVID-19 symptoms are characterized by systemic deterioration of the entire body, leading to significant physiological and functional imbalances. Common symptoms may be related to decreased short-term or long-term exercise capacity resulting from organ tissue damage, such as myocardial and pulmonary dysfunction. Currently, even vaccines and medications cannot effectively address the long-term consequences of COVID-19. Exercise training has been proven to improve exercise capacity and quality of life during the recovery period for various chronic disease patients.

A total of 24 patients will be included in the study. Following informed consent and baseline testing, the participants will be randomized in a 1:1 fashion to receive a 4-week aerobic exercise training or attention control.The main objective is to assess the effects of a 4-week aerobic exercise training program on cardiopulmonary fitness and long COVID-19 symptom improvement. Secondary objectives include: to characterize baseline and intervention-related changes in quality of life, depression, anxiety, insomnia status and perceived stress status.

ELIGIBILITY:
Inclusion Criteria:

1. 18-75 years old;
2. Complicated with at least one of the following symptoms within 3 months after COVID-19 infection, lasts for at least 2 months, and is not caused by other diseases: Cough, fatigue, memory loss, concentration problems, palpitation easily or rapid heartbeat, chest tightness or chest pain, pain (head, limbs, lower back), slow thinking or reaction, eye discomfort or decreased vision, shortness of breath or difficulty breathing at rest, diarrhea, loss of taste or decreased taste, insomnia, hair loss, other new symptoms after COVID-19 infection
3. Tested positive for COVID-19 quantitative Reverse Transcription-Polymerase Chain Reaction (RT-PCR) or antigen kit and turned negative for at least 4 weeks before inclusion;
4. The patient understands and signs the informed consent form.

Exclusion Criteria:

1. Infected with COVID-19 within one month
2. Conditions that may be worsened by exercise, such as acute cardiac insufficiency, exercise asthma, epilepsy, etc.
3. Physical disabilities caused by bone and joint or neuromuscular diseases,
4. Complicated with other serious diseases (such as unstable angina, resting oxygen saturation < 93%, untreated heart failure, uncontrolled arrhythmia, uncontrolled hypertension, uncontrolled type 2 diabetes),
5. Women during pregnancy and lactation;
6. Patients was assessed unsuitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-01-10 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Symptom improvement | Week 4
  Improvement or Recovery of Long-term COVID-19 Symptoms

SECONDARY OUTCOMES:
Peak oxygen uptake | Week 4
  The cardiopulmonary fitness assessed by Cardiopulmonary Exercise Test
Quality of life measured by 12-Item Short Form Health Survey (SF12) | Week 4
  Using 12-Item Short Form Health Survey to evaluate quality of life.
Anxiety measured by Generalized Anxiety Disorder 7-item scale (GAD-7) | Week 4
  Using Generalized Anxiety Disorder 7-item scale to evaluate anxiety status.
Depression measured by Patient Health Questionnaire 9-item scale (PHQ-9) | Week 4
  Using Patient Health Questionnaire 9-item scale to evaluate depression status.
Insomnia measured by Insomnia Severity Index (ISI) | Week 4
  Using Insomnia Severity Index to evaluate insomnia status.
Perceived stress measured by Perceived Stress Scale (PSS) | Week 4
  Using Perceived Stress Scale to evaluate stress level.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Crook H, Raza S, Nowell J, Young M, Edison P. Long covid-mechanisms, risk factors, and management. BMJ. 2021 Jul 26;374:n1648. doi: 10.1136/bmj.n1648. PMID 34312178
- [Background] Durstenfeld MS, Sun K, Tahir P, Peluso MJ, Deeks SG, Aras MA, Grandis DJ, Long CS, Beatty A, Hsue PY. Use of Cardiopulmonary Exercise Testing to Evaluate Long COVID-19 Symptoms in Adults: A Systematic Review and Meta-analysis. JAMA Netw Open. 2022 Oct 3;5(10):e2236057. doi: 10.1001/jamanetworkopen.2022.36057. PMID 36223120
- [Background] Longobardi I, Goessler K, de Oliveira Junior GN, Prado DMLD, Santos JVP, Meletti MM, de Andrade DCO, Gil S, Boza JASO, Lima FR, Gualano B, Roschel H. Effects of a 16-week home-based exercise training programme on health-related quality of life, functional capacity, and persistent symptoms in survivors of severe/critical COVID-19: a randomised controlled trial. Br J Sports Med. 2023 Oct;57(20):1295-1303. doi: 10.1136/bjsports-2022-106681. Epub 2023 May 10. PMID 37164620
- [Background] Jimeno-Almazan A, Franco-Lopez F, Buendia-Romero A, Martinez-Cava A, Sanchez-Agar JA, Sanchez-Alcaraz Martinez BJ, Courel-Ibanez J, Pallares JG. Rehabilitation for post-COVID-19 condition through a supervised exercise intervention: A randomized controlled trial. Scand J Med Sci Sports. 2022 Dec;32(12):1791-1801. doi: 10.1111/sms.14240. Epub 2022 Sep 23. PMID 36111386
- [Background] Josephson RA. Cardiac rehabilitation 2022. Prog Cardiovasc Dis. 2022 Jan-Feb;70:1. doi: 10.1016/j.pcad.2022.01.010. Epub 2022 Feb 1. No abstract available. PMID 35120977
- [Derived] Bai B, Xu M, Zhou H, Liao Y, Liu F, Liu Y, Yuan Y, Geng Q, Ma H. Effects of aerobic training on cardiopulmonary fitness in patients with long COVID-19: a randomized controlled trial. Trials. 2024 Oct 3;25(1):649. doi: 10.1186/s13063-024-08473-3. PMID 39363376
- See also: Clinical management of COVID-19: Living guideline — http://www.ncbi.nlm.nih.gov/books/NBK582435/
- See also: American College of Sports Medicine Guidelines for Exercise Testing and Prescription — https://books.google.co.uk/books/about/ACSM_s_Guidelines_for_Exercise_Testing_a.html?id=rpoMEAAAQBAJ&redir_esc=y